CLINICAL TRIAL: NCT06627036
Title: Dermoscopy vs. Standard Marking Practices for the Completeness of Excision of Keratinocyte Skin Cancers: a Single-centre Randomised Controlled Trial
Brief Title: Dermoscopy vs Standard Marking for the Completeness of Excision of Keratinocyte Skin Cancers: The ClearMark Trial
Acronym: ClearMark
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: To be confirmed
Record Dates: First submitted 2024-10-01; First posted 2024-10-04 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2024-10

CONDITIONS: Keratinocyte Skin Cancer
Keywords: Keratinocyte Cancer; Skin Cancer; Loupe magnification; Dermoscopy
MeSH Terms: conditions — Skin Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention - Dermoscopy (Experimental): Those allocated to this arm will have their suspicious skin lesion marked using a dermatoscope - a commercially available CE marked medical device used to magnify skin lesions and examine them with polarised light, in order to better characterise their borders and features
  Interventions: Device: Dermatoscope
- Control - Loupe magnification (No Intervention): Those allocated to this arm will have their suspicious skin lesion marked using the conventional method of surgical loupe magnification (2.5x - 3.5x) and theatre lights

INTERVENTIONS:
Device: Dermatoscope — For participants in the dermoscopy group, the marking will also be done preoperatively with a marker pen, but the lesion borders will be determined using a dermatoscope. A peripheral margin based on BAD guidelines will be marked similarly.
  Arms: Intervention - Dermoscopy

SUMMARY:
What is the study about? This study aims to improve the success rate of removal surgery for a common type of skin cancer. We will compare two different methods of marking (drawing where to remove) the skin before removing the lump: the normal method using magnifying glasses and theatre lights, and our proposed method using a handheld magnifying device called a dermatoscope.

Why is this study important? Skin cancer is the most common cancer in the UK. Currently, up to 10-11% of surgeries do not remove all of the cancer, which means patients may need more treatment. We do not know whether using a dermatoscope can help surgeons remove all of the cancer more often or not. If it does, it could prevent patients needing more surgery or time in hospital.

What will happen during the study? A computer will randomly allocate each participant to marking using the normal method, or using a dermatoscope. The surgery will then proceed as usual. After the surgery, patients will be asked to fill in a simple questionnaire about their thoughts. We will collect data from patients' notes to monitor the success of the surgery and any more treatments needed.

What will we measure? We will check participants records to see if the cancer was entirely removed. This is reported by a pathologist whenever a skin lump or bump is removed. In time, we will also look at 5-year recurrence of cancer, the need for additional treatments, any problems from the marking process, how happy patients are with the process, and the time it takes to perform the marking.

What is the pilot for? The study will need many hundreds of patients to pick up a meaningful result. Before we commit to recruiting this many people, we want to make sure that the way we run the study is acceptable. This means looking at the number of people we recruit each week, how easy it is to collect their data after their operation, and whether there are any areas that we can't use a dermatoscope, such as the curves around the eye, nose and ears. We will run the study in a smaller number of people (around 200) before deciding whether we can commit to recruiting everyone. This will also give us the chance to see whether we can run the study in more than one hospital.

DETAILED DESCRIPTION:
5 BACKGROUND AND RATIONALE 5.1.1 DESCRIPTION OF THE CONDITION Non-melanoma skin cancer (NMSC), also known as keratinocyte skin cancer (KSC), is the most prevalent cancer worldwide, particularly affecting fair-skinned individuals who lack protective skin pigment. In the United Kingdom (UK), the lifetime risk of developing keratinocyte skin cancer is 1 in 4 for men and 1 in 5 for women. The two primary types of keratinocyte cancer are basal cell carcinoma (BCC) and cutaneous squamous cell carcinoma (cSCC), accounting for approximately 80% and 20% of cases, respectively. Other rare types of skin cancer, such as Merkel cell carcinoma (MCC) and adenocarcinoma originating from skin gland cells, each constitute about 0.2% to 0.4% of all NMSCs.

BCCs generally develop after intense ultraviolet (UV) exposure during childhood and adolescence, whereas cSCCs are associated with cumulative UV exposure and chronic sun damage. The incidence of NMSC is rapidly increasing globally, with the UK experiencing an 8% annual rise. The incidence of cSCC appears to be growing faster than BCC, particularly among elderly men who have accumulated substantial sun damage over their lifetimes. This rise in incidence is primarily due to increased exposure to UV radiation, both from the sun and artificial sources like tanning beds.

Other significant risk factors for NMSC include advancing age, male gender, fair skin (Fitzpatrick types I and II), a history of skin cancer or severe sunburn, immunosuppression, family history of skin cancer, and exposure to carcinogens such as arsenic and ionizing radiation. However, the true incidence of NMSC is uncertain due to underreporting and inconsistencies in registration practices. In many countries, NMSCs are not always documented, and patients with multiple lesions may be registered only once, leading to a potential underestimation of the actual burden.

Despite their low mortality rates, NMSCs cause significant morbidity and represent a growing economic burden on healthcare systems worldwide (3). They frequently appear on the head and neck, where they can cause considerable local tissue destruction and disfigurement if treatment is inadequate or delayed. While BCCs are generally localized and rarely metastasize, cSCCs have the potential to spread to distant sites and become fatal.

The typical presentation of NMSC includes ulcers, nodules, or scaly patches that do not heal and continue to grow at varying rates. These lesions may bleed, itch, or cause significant local destruction. BCCs predominantly arise on the head, face, and neck, though some subtypes, such as superficial BCCs, are more common on the trunk and legs. Conversely, cSCCs typically occur on sun-exposed areas of the face, such as the ears, lips, and scalp, as well as on the neck, shins, and dorsum of the hands and forearms. However, both types can potentially develop anywhere on the body.

5.1.2 DESCRIPTION OF DIAGNOSIS AND MANAGEMENT Patients who present to primary care with a suspicious skin lesion should be referred either routinely for suspected BCC or urgently to a two-week wait clinic for suspected SCC or BCC when there is concern that delay might significantly impact the patient's prognosis. These patients undergo a thorough assessment by a specialist, either a dermatologist or a plastic surgeon. This assessment includes a focused history and clinical examination, dermoscopy, and medical photography. If the lesion is deemed suspicious, the patient is scheduled for a biopsy-either excisional or incisional-to establish a histological diagnosis. Management then depends on the biopsy results and, for SCCs, the TNM (Tumour, Node, Metastasis) staging, guided by the Local Skin Multidisciplinary Team (LSMDT) or the Specialist Skin Cancer Multidisciplinary Team (SSMDT).

A comprehensive history and meticulous clinical examination are crucial for the accurate diagnosis of referred skin lesions. Dermoscopy, widely used by dermatologists and plastic surgeons, is a non-invasive diagnostic tool for various skin lesions, including skin cancer. A dermatoscope is a handheld device that provides magnification from 10x to over 200x and has an adjustable built-in illumination system. By transilluminating the lesion, it visualises structures to the depth of the reticular dermis. Modern dermatoscopes achieve this without additional translucency-enhancing solutions by using polarised light, which filters out scattered light and allows visualisation of sub-stratal features. Dermoscopy helps discriminate between different skin lesions based on color, pattern, and structural analysis. When used by trained clinicians, dermoscopy significantly improves the accuracy of skin cancer diagnosis for both melanoma and keratinocyte cancers. It increases sensitivity for skin cancer detection, decreases the benign-to-malignant biopsy ratio, identifies cancers at an earlier stage, and allows for the diagnosis of different BCC subtypes compared to naked eye examination (NEE). Dermatoscopic characteristics of lesions show good correlation with histopathological features of skin lesions, making dermoscopy an invaluable part of the diagnostic approach to suspicious skin lesions.

Once a lesion is inspected and deemed suspicious for skin cancer, a biopsy is offered to confirm the diagnosis and assess risk. The first-line treatment is often an excision biopsy, where the entire lesion is removed with a margin of normal-appearing skin. This approach aims to achieve complete excision and treatment without the need for further surgery or treatment. Other biopsy options include incisional, punch, and shave biopsies, which provide a smaller sample of the lesion for histopathological analysis. Reconstruction, if needed, can be immediate or delayed, based on the clarity of the clinical margins.

The BAD has published guidelines based on studies using Mohs micrographic surgery (MMS) regarding recommended peripheral skin margins for BCCs and SCCs, depending on clinical and pathological criteria that classify them as low, high, or very high (only for SCCs) risk. For BCCs, the recommended margins are 4-5mm for low-risk lesions and 5-10mm for high-risk lesions. For SCCs, the recommended margins are ≥4mm for low-risk, ≥6mm for high-risk, and ≥10mm for very high-risk lesions. These margins are assessed preoperatively, typically using theatre lights and loupe magnification, as per BAD recommendations.

Other treatment options include Mohs micrographic surgery, especially for recurrent or poorly defined lesions in cosmetically sensitive areas, electrodessication and curettage (EDC), cryosurgery, radiotherapy (RT), photodynamic therapy (PDT), topical chemotherapy (e.g., 5-fluorouracil), and topical immunotherapy (e.g., imiquimod). Non-surgical methods lack histological confirmation of tumor clearance and are typically reserved for low-risk lesions, with the exception of RT, which is used routinely for older adults (≥60) with lesions of any risk category in well-vascularised anatomical sites who decline or are unsuitable for surgery.

5.1.3 RATIONALE Skin cancer is the most prevalent cancer in the UK, with a lifetime risk of 1 in 4 for men and 1 in 5 for women, and an annual incidence increase of 8%. The primary treatment approach involves complete surgical excision, with UK dermatologists alone performing approximately 200,000 NMSC excisions annually. However, incomplete excision rates vary, ranging from 9% for squamous cell carcinomas to 11% for basal cell carcinomas. This could mean up to 20,000 patients annually that are inadequately treated. Incomplete excision exacerbates morbidity, imposing additional burdens such as the need for further surgeries or radiotherapy, psychological distress, productivity loss, and increased costs for the NHS (National Health Service). These costs encompass theatre utilisation, dressing materials, consultant-led clinic appointments, and prolonging already stretched waiting lists.

The British Association of Dermatologists suggests a 95% complete excision rate as the gold standard when adhering to their guidelines for surgical marking, indicating ample room for enhancement. One way of potentially improving the rate of incomplete excision is by marking the lesion pre-excision with a dermatoscope - a handheld device providing high-factor magnification and polarised and non-polarised light specifically designed for the assessment of skin lesions. Although dermoscopic marking of tumour margins shows promise, evidence remains sparse. Furthermore, the use of dermoscopy for surgical margins vs. common practices with theatre lights and loupes has not been formally compared with robust and high-quality prospective studies. We are therefore proposing a study to evaluate the effectiveness of using dermoscopy for lesion marking, prior to lesion excision. Notably, our inquiry has been identified as the second most crucial research question in skin cancer surgery by a James Lind Alliance (JLA) Priority Setting Partnership (PSP). By comparing standard practices, using loupes and theatre lights, with dermoscopy for preoperative marking of skin lesions we will therefore specifically help to address the PSP priority of "What is the most effective way of determining the borders of the skin cancer before skin cancer surgery?".

5.1.4 OBJECTIVES To conduct a single-centre randomised controlled trial (RCT) comparing dermoscopy-guided excision with loupe-magnified excision in patients undergoing suspected keratinocyte cancer excision

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older who are scheduled for the excision of a suspected non-melanoma skin cancer lesion as part of a day-case surgery list at Hull University Teaching Hospitals are eligible for inclusion in the study.

Exclusion Criteria:

* Lesions that are inaccessible to dermoscopic assessment due to anatomical locations or conditions that prevent effective use of the dermatoscope.
* Lesions that are determined to be benign or pigmented upon initial evaluation and therefore do not meet the criteria for suspected keratinocyte skin cancer.
* Lesions scheduled for incisional, punch, or shave biopsy procedures, as these methods do not provide complete peripheral margin clearance.
* Lesions that are histologically confirmed as benign following excision and examination by a pathologist.
* Patients who decline to participate in the study.
* Patients who are unable to provide informed consent due to a lack of mental capacity or other reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1376 (Estimated)
Dates: Start 2024-11-21 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2031-05-31 (Estimated)

PRIMARY OUTCOMES:
Excision completeness at the lateral margin | Measured on histology reports available 6 weeks post-operatively
  The primary outcome will assess the completeness of excision at the peripheral margin, confirmed by histological examination of the skin lesion, for patients undergoing excision biopsy of suspected keratinocyte skin cancer. As dermoscopy can only assess up to the depth of the reticular dermis, the completeness of excision at the deep margin will not be evaluated in this study.

SECONDARY OUTCOMES:
5 Year Recurrence Rate | 5 years
  We will measure recurrence of the skin lesion within 5 years of lesion excision
5 Year additional treatment rate | 5 years
  We will measure additional treatment for the index lesion within 5 years of lesion excision - this includes wider surgical excision, radiotherapy, cryotherapy, electrochemotherapy, and immunotherapy
Adverse Events relating to lesion marking | During the time of the procedure and for up to 3 hours post-operatively
  We will collect data on adverse events relating only to the lesion marking procedure
Patient acceptability and satisfaction | During the time of procedure, measured within 1 hour of the end of the surgical procedure
  We will measure patient satisfaction on a 1-10 visual analogue scale, with 1 being completely unacceptable and 10 being completely acceptable
Time required for marking | The interval from the patient entering the theatre to knife-to-skin
  We will measure the time required for marking with each method (measured in minutes using operative records, defined as the interval from the patient entering the theatre to knife-to-skin).

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Totty, MBBS MRCS PGCert MD(Res) FHEA, Principal Investigator — Hull York Medical School
Locations (1):
- Castle Hill Hospital, Hull, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
In the interests of open science, the study protocol and approved documents will be made available via the open science framework (OSF) website. A shortened protocol will be prepared for publication in a peer reviewed journal. Once collected, fully anonymised data will be made available using the open science framework, along with any statistical code used for the analysis of the data.
Supporting Information: Study Protocol
Time Frame: IPD will be available for the duration of the study and for up to 3 years following publication in a peer reviewed journal.